CLINICAL TRIAL: NCT01442818
Title: Patient Satisfaction and Pain Control Following Reconstructive Vaginal Surgery: A Randomized Trial Comparing Patient-Controlled Intravenous Analgesia (PCA) to Scheduled Intravenous Analgesia
Brief Title: Patient Satisfaction and Pain Control Following Reconstructive Vaginal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10072
Record Dates: First submitted 2010-09-08; First posted 2011-09-29 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Post Operative Pain
Keywords: vaginal reconstructive surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Scheduled IV post op (Experimental): Patient's will receive scheduled nurse administered IV pain medications post operatively.
  Interventions: Drug: Dilaudid IV Scheduled
- PCA post op (Experimental): Patients will receive PCA for pain control post operatively.
  Interventions: Drug: Dilaudid PCA

INTERVENTIONS:
Drug: Dilaudid PCA — PCA setting of 0.3mg demand dose, 8 minute lock out interval, and 5mg 4-hour limit.
  Other Names: hydromorphone
  Arms: PCA post op
Drug: Dilaudid IV Scheduled — Nurse administered IV Dilaudid 0.5mg every 2 hours.
  Other Names: hydromorphone
  Arms: Scheduled IV post op

SUMMARY:
The investigators hypothesize that patient controlled analgesia (PCA) provides superior pain relief and patient satisfaction when compared to scheduled intravenous analgesia following vaginal reconstructive surgery.

DETAILED DESCRIPTION:
The investigators hypothesize that patient controlled analgesia (PCA) provides superior pain relief and patient satisfaction when compared to scheduled intravenous analgesia following vaginal reconstructive surgery.

In order to determine if there is a significant correlation, secondary outcomes will include the daily and total narcotic volume used, common side effects from the opioid including nausea, vomiting, or pruritis, length of hospital stay, timing of flatus and first bowel movement, all complications, and procedure performed.

ELIGIBILITY:
Inclusion Criteria:

* The patients will be limited to those from the Division of Urogynecology to ensure similar surgical techniques. They will be between the ages of 18 and 70 and undergoing major vaginal reconstruction.
* All patients must undergo vaginal reconstructive surgery including: anterior repair, posterior repair, and intraperitoneal vaginal vault suspension. The addition of vaginal hysterectomy, enterocele repair, or suburethral sling is not cause for exclusion.

Exclusion Criteria:

* Any patient who has an allergy to hydromorphone/Dilaudid.
* Any patient already taking chronic opioids, defined as daily use.
* All patients with renal insufficiency or failure.
* All patients with liver failure.
* Any patient who is not having general anesthesia.
* Any patient undergoing abdominal or laparoscopic procedures: sacral colpopexy, laparoscopic hysterectomy or oophorectomy, Burch procedure, or any procedure that enters the abdominal fascia.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Patient Pain Control | post operative day 1
  Patient's reported pain on a VAS on all postoperative day one.

SECONDARY OUTCOMES:
Patient Satisfaction with Pain Control | post operative day 1
  Patient's satisfaction with pain control on a VAS on all postoperative day one.
patient perceived pain at 2 weeks | 2 weeks post op
  VAS for pain will be filled out at the patient's two week post op office visit.
patient dissatisfaction with pain control at 2 weeks | 2 weeks post op
  patient will fill out a VAS for satisfaction with pain control at their two week post operative visit.

CONTACTS AND LOCATIONS:
Overall Officials: Catrina C Crisp, MD, Principal Investigator — TriHealth Division of Urogynecology
Locations (1):
- Good Samaritan Hospital, Cincinnati, Ohio, United States